CLINICAL TRIAL: NCT03925857
Title: Prevention of Sepsis-related Organ Dysfunction With Allocetra-OTS
Acronym: P-SOFA-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enlivex Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: ENX-CL-02-001; MOH_2019-02-17_005970 (Registry Identifier: Israeli Ministry of Health)
Record Dates: First submitted 2019-04-01; First posted 2019-04-24 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Organ Dysfunction Syndrome Sepsis
Keywords: Allocetra-OTS; Cell based therapy; Apoptotic cells
MeSH Terms: conditions — Toxemia

STUDY DESIGN:
Intervention Model Description: One Dose: 3 Sepsis patients will be treated with Allocetra-OTS, following safety assessment additional 3 patients will be treated (total 6 patients).
  Two doses: Once safety is established 4 sepsis patients will be treated with 2 doses of Allocetra-OTS; The first, as in the first six patients and the second 48 hr following the first treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allocetra-OTS (Experimental): Standard of Care (SOC) Drug: One dose Allocetra-OTS 140 140x106 /kg
  Interventions: Biological: Allocetra-OTS
- Allocetra-OTS Two doses (Experimental): Standard of Care (SOC) Drug: Two doses Allocetra-OTS 140 140x106 /kg
  Interventions: Biological: Allocetra-OTS

INTERVENTIONS:
Biological: Allocetra-OTS — Allocetra-OTS contains allogeneic donor mononuclear enriched cells in the form of a liquid suspension with at least 40% early apoptotic cells. The suspension is prepared with Ringer's lactate solution.

SUMMARY:
The trial evaluates the safety and efficacy of one and two doses of the study drug, Allocetra-OTS, in patients who have been diagnosed with sepsis.

DETAILED DESCRIPTION:
The study drug, Allocetra-OTS is a cell-based therapeutic composed of donor apoptotic cells. The product contains allogeneic mononuclear enriched cells in the form of a liquid suspension with at least 40% early apoptotic cells. The study drug, Allocetra-OTS, is based on the known activity of apoptotic cells to contribute to maintenance of peripheral immune homeostasis. As altered immune response is associated with organ dysfunction in sepsis, the possibility is being tested that the study drug can improve the condition of sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Suspected, presumed or documented infection from any source.
* Initiation of antibiotics.
* Meets Sepsis 3 criteria: The presence of organ dysfunction as identified by a total SOFA score ≥ 2 points above baseline.
* Adult male or female, age between 18 and 85.
* GCS of >13 with verbal score of 5.
* Signed written informed consent by the patient.

Exclusion Criteria:

* Participation in an interventional investigational trial within 30 days prior to diagnosis of sepsis.
* Significant trauma requiring hospitalization within 30 days prior to diagnosis of sepsis.
* Surgical intervention or hospitalization within 45 days prior to diagnosis of sepsis.
* Pregnancy or breast-feeding female.
* Progressive or poorly-controlled malignancies or < 6 month after active treatment for cancer (chemotherapy or irradiation).
* Terminally ill patients defined as patients that prior to the current hospitalization are expected to live < 6 months (as assessed by the physician responsible for the patient).
* Known active acute or chronic viral infections, e.g. Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV) or other chronic infection.
* Known severe chronic respiratory health problems with severe pulmonary hypertension (≥40 mmHg) or respirator dependency.
* Known active upper gastrointestinal (GI) tract ulceration or hepatic dysfunction including but not limited to: biopsy-proven cirrhosis; portal hypertension; episodes of past upper GI bleeding attributed to portal hypertension; or prior episodes of hepatic failure, encephalopathy, or coma.
* Known New York Heart Association (NYHA) class IV heart failure or unstable angina, ventricular arrhythmias, active ischemic heart disease, or myocardial infarction within six months prior to diagnosis of sepsis.
* Known immunocompromised state or medications known to be immunosuppressive.
* Organ allograft or previous history of stem cell transplantation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-27 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-01-12 (Actual)

PRIMARY OUTCOMES:
Assessment of safety by determining the number of participants with any Adverse Events (AE),Serious Adverse Events (SAE) and fatal SAE | 28 days follow up
  Incidence rates of any Adverse Events (AE), Serious Adverse Events (SAE) and fatal SAE

SECONDARY OUTCOMES:
Organ function or support measurements | 28 days follow up
  * Ventilator-free days, and/or
  * Vasopressor-free days, and/or
  * Days without renal replacement therapy (dialysis) and/or days with creatinine ≤ baseline +20%, and/or
  * Days with ≥ 100x109/L platelets count, and/or
  * Days with ≤ three times normal ALT (Alanine transaminase) and AST ••(Aspartate Aminotransferase) levels and/or ≤ two times normal bilirubin levels and/or
  * Days with return to GCS (Glasgow Coma Scale) 15
Mortality | 28 days follow up
  Incidence rate of Moratlity from any cause
Hospitalization | 28 days follow up
  Cumulative days in Intensive care unit (ICU) or Intermediate Care Units (IMU) and/or in hospital.
CRP | 28 days follow up
  Time to C-reactive protein (CRP) < 20 mg/L.
Lactate levels | 28 days follow up
  Time to normal + 20% lactate levels

CONTACTS AND LOCATIONS:
Overall Officials: Dror Mevorach, Prof, Study Director — Enlivex Therapeutics LTD Email:mevorachd@gmail.com
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Heerden PV, Abutbul A, Sviri S, Zlotnick E, Nama A, Zimro S, El-Amore R, Shabat Y, Reicher B, Falah B, Mevorach D. Apoptotic Cells for Therapeutic Use in Cytokine Storm Associated With Sepsis- A Phase Ib Clinical Trial. Front Immunol. 2021 Sep 30;12:718191. doi: 10.3389/fimmu.2021.718191. eCollection 2021. PMID 34659208